CLINICAL TRIAL: NCT05527704
Title: a Multicentre, Double-blind, Randomized, Placebo-controlled Phase III Trial of the Inhaled β2-adrenergic Receptor Agonist Salbutamol for Transient Tachypnoea of the Newborn (the REFSAL Trial)
Brief Title: the Inhaled β2-adrenergic Receptor Agonist for Transient Tachypnoea of the Newborn (the REFSAL Trial)
Acronym: REFSAL
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Collaborators: University of Ottawa (Other); Jagiellonian University (Other); Pomeranian Medical University Szczecin (Other); Poznan University of Medical Sciences (Other); Jan Biziel University Hospital No 2 in Bydgoszcz (Other); Neonatology Unit, Specialist Hospital No 2, Bytom (Unknown); University of Rzeszow (Other); University in Zielona Góra (Other); SZPITAL SPECJALISTYCZNY IM. ŚW. RODZINY w Warszawie (Unknown); Neonatology Unit, Szpital Specjalistyczny Pro-Familia, Rzeszow (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019/ABM/01/00058/P/03; 2020-003913-36 (EudraCT Number)
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-09

CONDITIONS: TTN; Respiratory Failure; PPHN
Keywords: TTN; PPHN; CPAP; Salbutamol
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CPAP+Salbutamol (Active Comparator): All patients will receive nCPAP at 5-6 cm H2O pressure with an oxygen concentration of 21% or more to maintain preductal saturation between 90% and 95%. Patients assigned to the active group will be treated with 0.15 mg/kg body weight (diluted in 3 mL 0.9% NaCl) nebulised salbutamol (Ventolin®, GlaxoSmithKline, Dublin, Ireland) for 30 min.
  Interventions: Drug: Salbutamol
- CPAP+Placebo (Placebo Comparator): Patients in the placebo group will also receive nCPAP at 5-6 cm H2O pressure with an oxygen concentration of 21% or more to maintain preductal saturation between 90% and 95%. In addition, patients will receive 3 mL nebulised 0.9% NaCl administered for 30 min. as a placebo
  Interventions: Drug: 0,9% Chloride Sodium

INTERVENTIONS:
Drug: Salbutamol — Patients assigned to the active group will be treated with 0.15 mg/kg body weight (diluted in 3 mL 0.9% NaCl) nebulized salbutamol (Ventolin®, GlaxoSmithKline, Dublin, Ireland) for 30 min.
  Other Names: Albuterol
  Arms: CPAP+Salbutamol
Drug: 0,9% Chloride Sodium — 3 mL nebulized 0.9% NaCl administered for 30 min.
  Other Names: 0,9% NaCl
  Arms: CPAP+Placebo

SUMMARY:
Clinical trial evaluating the efficacy and safety of salbutamol for the treatment of neonates with a gestational age between 32 and 42 weeks with transient tachypnoea of the newborn (TTN).

DETAILED DESCRIPTION:
Multicentre, double-blind, phase III trial will include infants with a gestational age between 32 and 42 weeks and respiratory disorders treated in neonatal intensive care units in Poland. Infants will be enrolled no later than 24 h after birth and will be randomly assigned (1:1) to receive nebulized salbutamol with nCPAP or placebo (nebulized 0.9% NaCl) with nCPAP. The primary outcome is the percentage of infants with TTN who develop PPHN.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age at birth between 32 and 42 weeks.
2. Respiratory disorders (tachypnea and expiratory grunting) lasting longer than 15 minutes after birth, or present for at least 15 minutes in the first six hrs of life, or a need for non-invasive respiratory support between birth and six hrs of life.
3. Available chest radiographs obtained within six hrs after birth.
4. Available parameters of the acid-base balance (blood pH, partial pressure of O2 and CO2, base excess) and blood serum ionogram for Na+, K+, Ca2+ evaluated in the umbilical cord blood sample.

Exclusion Criteria:

1. Need for intubation directly after birth or perinatal asphyxia, defined as abnormal acid-base parameters detected in an umbilical cord blood sample (pH <7.0 or base excess < -14 mmol/L).
2. Multiple apnea-brady that require immediate intubation before a trial of NIV
3. Age >24 h.
4. Meconium aspiration syndrome.
5. Air leak syndrome.
6. Congenital heart disease.
7. Congenital diaphragmatic hernia.
8. Other severe congenital malformations and genetic disorders (diagnosed before and after birth) associated with increased risk of respiratory failure.
9. The need for a surfactant administration immediately after birth, regardless of the method of its administration (respiratory distress syndrome - RDS)

Max Age: 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 608 (Estimated)
Dates: Start 2021-12-31 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Persistent Pulmonary Hypertension of the Newborn (PPHN) | 7 days of life
  PPHN defined as the need for ventilation with FiO2 >0.30 and features of increased pulmonary pressure on echocardiogram

SECONDARY OUTCOMES:
the severity of respiratory distress | 48 hrs of life
  assessed with the modified TTN Silverman score
need for intubation | 7 days of life
  frequency of need for intubation
duration of ventilation | 7 days of life
  duration of ventilation e.g. non-invasive ventilation
duration of hospitalization | up to first month of life
  duration of hospitalisation after birth

CONTACTS AND LOCATIONS:
Overall Officials: Renata Bokiniec, MD, PhD, Principal Investigator — Medical University of Warsaw
Locations (1):
- Medical University of Warsaw, Warsaw, Poland

REFERENCES:
- [Derived] Madajczak D, Daboval T, Lauterbach R, Loniewska B, Blaz W, Szczapa T, Sadowska-Krawczenko I, Michalak-Kloc M, Slawska H, Borszewska-Kornacka M, Bokiniec R; REFSAL Study Group. Protocol for a multicenter, double-blind, randomized, placebo-controlled phase III trial of the inhaled beta2-adrenergic receptor agonist salbutamol for transient tachypnea of the newborn (the REFSAL trial). Front Pediatr. 2023 Jan 12;10:1060843. doi: 10.3389/fped.2022.1060843. eCollection 2022. PMID 36714639